CLINICAL TRIAL: NCT04592562
Title: Genicular Artery Embolization to Reduce Pain Associated With Unilateral Mild to Moderate Osteoarthritis: A Pilot Study to Assess Feasibility
Brief Title: Genicular Artery Embolization to Reduce Pain Associated With Unilateral Mild to Moderate Osteoarthritis
Acronym: GAE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: IRB20-0868
Record Dates: First submitted 2020-10-14; First posted 2020-10-19 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-05

CONDITIONS: Knee Osteoarthritis
Keywords: Genicular Artery Embolization; Knee Pain; Knee Osteoarthritis; Genicular Artery; Embolization; Pain Management
MeSH Terms: conditions — Osteoarthritis, Knee; Agnosia

STUDY DESIGN:
Intervention Model Description: Patients who meet study eligibility will undergo the novel Genicular artery embolization procedure by a licensed Interventional Radiologist at the University of Chicago Medical Center.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- GAE Arm (Experimental): Patients who meet study eligibility will be scheduled to undergo the Genicular Artery Embolization procedure and will subsequent be followed for 12 months after their procedure.
  Interventions: Device: the Terumo Hydropearl® microspheres device

INTERVENTIONS:
Device: the Terumo Hydropearl® microspheres device — Genicular artery embolization (GAE) is a new, minimally invasive investigational not yet approved therapy. In previous studies, this procedure has provided pain relief in patients with mild to moderate OA in the short to midterm. We will be utilizing the Terumo Hydropearl® microspheres particle beads during the GAE procedures. The procedure will take place utilizing fluoroscopic and ultrasound guidance. Following catheterization of the femoral artery, angiography of the affected limb will be performed to define the genicular arterial anatomy. Genicular arteries demonstrating abnormal vascularity and corresponding to the site of the patient's pain will be catheterized and embolized using microspheres. Prior to and after embolization, parametric imaging will be performed utilizing proprietary software to quantify changes in blood flow to the target area
  The intended use of the Terumo Hydropearl® microspheres device is to embolize the geniculate artery branch.

SUMMARY:
The goal of this study is to perform a feasibility study to show the effectiveness of the genicular artery embolization procedure in reducing bilateral or unilateral osteoarthritic knee pain at 12 months as measured by WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) score, Knee Injury and Osteoarthritis Outcome (KOOS) score, and Oswestry Disability Index.

DETAILED DESCRIPTION:
This is a single-center, pilot study to assess the feasibility of a study show the effectiveness of the genicular artery embolization (GAE) in reducing arthritic pain and dysfunction associated with mild to moderate Bilateral or unilateral osteoarthritis of the knee. Patients with bilateral or unilateral Grade 1-3 Osteoarthritis as diagnosed on standing weight-bearing knee radiographs per the Kellen-Lawrence Grading scale, will be offered enrollment to the study. Following a screening questionnaire, these patients will then be enrolled in this study. Baseline MRI will be obtained prior to the GAE procedure. Follow up intervals will include 3, 6, 9, and 12 months with the primary objective measured by a clinician as the WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) score, Knee Injury and Osteoarthritis Outcome (KOOS) score, and Oswestry Disability Index at the 12-month follow up visit. Patients will also undergo 1 year follow up MRI to be interpreted by a diagnostic radiologist with subspecialty training in musculoskeletal radiology. This radiologist will compare the treated knee to the baseline screening according to the WORMS classification (Whole Organ Magnetic Resonance Scoring) to assess for radiologic changes of osteoarthritis and any adverse effects.

ELIGIBILITY:
Inclusion Criteria:

We intend to include patients who meet the following criteria in the study:

1. Patients aged 40-80
2. Bilateral or Unilateral knee pain attributed to osteoarthritis
3. Grade 1-3 Osteoarthritis as diagnosed on standing weight-bearing knee radiographs per the Kellen-Lawrence Grading scale
4. Knee pain >6 months refractory to conservative medical management (NSAIDs, paracetamol, intra-articular injections, physiotherapy/exercise, weight loss, etc.)

Exclusion Criteria:

* We plan to exclude patients who meet any of the following criteria:

  1. Active malignancy
  2. Active infection of the affected knee
  3. Platelets <50,000
  4. INR >1.8 (unless on anticoagulation that can be reversed)
  5. Corticosteroid injection of the affected knee within 3 months
  6. Rheumatoid arthritis or other seronegative arthropathy
  7. Previous surgery (excluding arthroscopy) of the affected knee
  8. Grade 4 per Kellgren-Lawrence Grading Scale of the affected knee
  9. Pregnancy or expected pregnancy
  10. GFR <30
  11. Anaphylactic reaction to iodinated contrast
  12. Moderate to severe pain in other lower limb joints
  13. Body weight >400 lbs. (Procedure table weight limit)
  14. BMI >50
  15. Patients at high risk for contrast nephropathy

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-05-28 (Actual)

PRIMARY OUTCOMES:
WOMAC Scale | 12 Months
  The reduction of Bilateral or unilateral knee pain and dysfunction associated with mild to moderate osteoarthritis at 12 months as measured by WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) score
KOOS Scale | 12 Months
  The reduction of Bilateral or unilateral knee pain and dysfunction associated with mild to moderate osteoarthritis at 12 months as measured by the Knee Injury and Osteoarthritis Outcome (KOOS) score
Oswestry Disability Index | 12 Months
  The reduction of Bilateral or unilateral knee pain and dysfunction associated with mild to moderate osteoarthritis at 12 months as measured by the Oswestry Disability Index

SECONDARY OUTCOMES:
WOMAC for Knee Pain and Dysfunction | 12 Months
  To assess reduction in knee pain and dysfunction at 3, 6, and 9-months for subjects undergoing the GAE procedure using the WOMAC scale
KOOS for Knee Pain and Dysfunction | 12 Months
  To assess reduction in knee pain and dysfunction at 3, 6, and 9-months for subjects undergoing the GAE procedure using the KOOS scale
Oswestry Disability Index for Knee Pain and Dysfunction | 12 Months
  To assess reduction in knee pain and dysfunction at 3, 6, and 9-months for subjects undergoing the GAE procedure using the Oswestry Disability Index
VAS for Pain | 12 Months
  To report the outcomes of Visual Analog Score (VAS) for pain at 0, 3, 6, 9, and 12 months post.
Six-Minute Walk Test for Functional Improvement | 12 months
  To determine and report six-minute walk test performance and to assess functional improvement at baseline, 3, 6, 9, and 12 months
Thirty-Second Chair Test for Performance | 12 Months
  To determine and report thirty-second chair stand test performances and to assess functional improvement at baseline, 3, 6, 9, and 12 months.
Opiate Usage | 12 Months
  Change in usage of opiate or opiate-equivalent medications calculated by using the internal opioid change log, kept and updated by the study team from baseline to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Osmanuddin Ahmed, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No